CLINICAL TRIAL: NCT04694794
Title: D-CRSE: Diminish Chemotherapy Related Side Effects Through Patient Education in Patients With Breast OR Gastrointestinal Cancer Who Are Undergoing Cytotoxic Chemotherapy
Brief Title: Diminish Chemotherapy Related Side Effects Through Patient Education
Acronym: D-CRSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Monali Vasekar, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PSCI-19-112
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Chemotherapeutic Toxicity; Chemotherapeutic Agent Toxicity; Chemotherapy Effect

STUDY DESIGN:
Intervention Model Description: Single arm interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Single arm, interventional. All participants will be administered Educational Brochure to educate them regarding management of side effects experienced during chemotherapy treatment
  Interventions: Other: Educational Brochure

INTERVENTIONS:
Other: Educational Brochure — Participants will be provided with Education Brochure developed by the study team to provide information to patients about managing side effects related to chemotherapy

SUMMARY:
Currently, there is a lack of patient education materials regarding cytotoxic chemotherapy side effects, research supported treatments, and the utilization of CAM by cancer patients at Penn State Cancer Institute. The investigators aim to develop an educational brochure, which educates patients about the chemotherapy side effects they may experience, and provide them with the tools to address the problem themselves, know when to contact their medical oncologist, and understand when it is appropriate to go to the Emergency Department. By educating patients regarding these problems, patient anxiety may decrease, the number of calls into the oncologist office may decrease, and Emergency Department visits may decrease, which would decrease costs for the patient, the hospital, and the health system. If this intervention is found to be useful and impactful, it can be further utilized within the Cancer Institute by other disease teams, by other Penn State institutions, or by other institutions across the country.

DETAILED DESCRIPTION:
The diagnosis of cancer is a life-altering event which can cause a large amount of distress in patients. One of the several factors that impacts a patient's level of distress, is their fear of the diagnosis and their lack of information in the beginning their cancer journey. Understandably, many patients turn to easily accessible but disreputable resources, such as the internet, to learn and mentally prepare themselves for this journey. Friends and family members may also provide advice or recommendations which may not always be scientifically supported. Disreputable resources often have incorrect information that can scare or mislead a patient, which can severely impact their health and fight against cancer. In order to help patients fight these fears and become properly equipped for the cancer journey, care teams must address the education of patients, especially the education about the chemotherapy treatment process and potential side effects.

The primary purpose of this pilot study is to determine the utility of a brochure to educate breast and gastrointestinal cancer patients undergoing cytotoxic chemotherapy about the side effects of treatment, in addition to providing them with tools and recommendations to lessen the impact of these side effects on their quality of life. A questionnaire-based approach and the Patient Education Material Assessment Tool (PEMAT) will be employed to evaluate participant's responses in a variety of domains, such as understandability, actionability, and utility of the brochure. The Memorial Symptom Assessment Scale (MSAS) will be used to capture the specific chemotherapy side effects that each patient is experiencing throughout their treatment. Emotional Thermometer Scales (ETS) will be utilized to assess patients' feelings of depression, anxiety, anger, and distress at the beginning and end of their treatment. Survey questions will be utilized at interval time points (baseline plus 6 and 12 weeks) to evaluate the overall impact of the brochure on their quality of life and symptom management. All patients will receive the brochure and fill out the associated assessment scales and tools. The investigator's hypothesis is that a brochure providing information and tools to address the side effects of breast and gastrointestinal cancer cytotoxic chemotherapy will have utility in cancer clinics and allow patients to improve their quality of life by following the scientifically supported recommendations within the brochure.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of breast or gastrointestinal cancer, at any stage or progression, who are cytotoxic chemotherapy treatment naïve and initiating treatment or have newly begun cytotoxic chemotherapy within the last 6 weeks. Patients receiving multiple therapy forms, such as immune or humoral, can be included if they are also receiving cytotoxic chemotherapy as a part of their regimen. All patients will receive the brochure, therefore, there will not be a control arm in this study.

  1. Adult >20 year of age
  2. Ability to understand and read written English without any functional difficulty
  3. ECOG performance status 0-3
  4. May be involved with other cancer trials being offered at the Penn State Cancer Institute

Exclusion Criteria

1. Inability to give informed consent
2. Pregnant females
3. Inability to understand or read written English
4. Patients who have previously undergone cytotoxic chemotherapy at any point in their lifetime or began chemotherapy for their breast or gastrointestinal cancer greater than 6 weeks from the initiation of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Utility of Educational Brochure assessment | 12 weeks
  • Assessment of the utility of a brochure which educates breast and gastrointestinal cancer patients about the potential side effects of cytotoxic chemotherapy, as measured by the validated PEMAT survey score mean and standard deviation from baseline compared to 6 and 12 weeks post baseline assessment.
  The Patient Education Materials Assessment Tool for Printable Materials (PEMAT-P) scale used for above outcome ranges from minimum of score 0 percent to maximum score of 100 percent. Higher values indicate better outcome.

SECONDARY OUTCOMES:
Symptom Assessment | 12 weeks
  • Assessment of participant symptoms during cytotoxic chemotherapy treatment utilizing the MSAS.
  Memorial Symptom Assessment Scale used for above outcome ranges from minimum of score 0 to maximum score of 364. Higher values indicate presence of more and severe symptoms thus indicating worse outcome.
Emotional Assessment | 12 weeks
  • Assessment of participant emotions at the beginning and end of the study by comparing ETS scores.
  The Emotional Thermometer Scale used for above outcome ranges from minimum of score 0 to maximum score of 50. Higher values indicate presence of more and severe symptoms thus indicating worse outcome.
Baseline Educational Assessment | Baseline
  • Identification of participants with immediate family member (child, spouse, parent) who underwent cytotoxic chemotherapy and participant's education level through questionnaire.

OTHER OUTCOMES:
Feasibility Assessment | 12 weeks
  • Measure of participant withdraw rate from study as a representation of feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Monali Vasekar, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Information will be collected in De identified manner . IPD will not be shared with any other researchers.